CLINICAL TRIAL: NCT06418373
Title: Development and Polit Study of an Intervention Program to Enhance the Transition Readiness of Adolescents With Congenital Heart Disease
Brief Title: Development and Polit Study of Get Ready With my Heart Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHFudanU0505
Record Dates: First submitted 2024-05-06; First posted 2024-05-17 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Transition to Adult Care; Congenital Heart Disease
Keywords: Transition to adult care; CHD; Adolescent
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional intervention group (Active Comparator): Based on the current congenital heart disease care standards at Fudan University Children's Hospital, health education and medical management for adolescent CHD
  Interventions: Behavioral: Conventional intervention
- Intervention group (Experimental): Patients and their caregivers implement the "Get Ready with My Heart Program"
  Interventions: Behavioral: Get Ready with My Heart Program; Behavioral: Conventional intervention

INTERVENTIONS:
Behavioral: Get Ready with My Heart Program — In the intervention group, adolescent CHD patients undergo a comprehensive assessment by cardiology and cardiothoracic experts to determine their suitability for transitional care management. Based on the "Get Ready with My Heart Program," a personalized transition plan is developed, offering courses and resources that enhance self-management skills such as medication management, symptom monitoring, and health record maintenance. Throughout the transition period, regular support and follow-ups are provided to ensure that both patients and their families are adequately supported. The program includes regular assessments of transition readiness and quality of life changes to understand the intervention's impact and make necessary adjustments. Additionally, feedback is actively collected from patients and their families to continuously improve and refine the program.
  Arms: Intervention group
Behavioral: Conventional intervention — Adolescent CHD patients and their caregivers receive comprehensive health education and medical management. Upon admission, a detailed assessment of each patient's medical history and physical examination is conducted. A treatment and perioperative care plan is then tailored, including medication management with anticoagulants and antiarrhythmics, and surgery-related health guidance. Regular cardiac monitoring and follow-up assessments ensure treatment effectiveness and health status updates. Post-discharge, patients receive lifestyle management advice through remote consultations, focusing on diet and physical activity. Additionally, training on recognizing and managing emergencies is provided, equipping patients and caregivers to handle potential crises effectively. This holistic approach aims to improve both immediate and long-term health outcomes for adolescent CHD patients.

SUMMARY:
The goal of this clinical trial is to learn if the Get Ready with my Heart Program developed based on SMART theory is applicable for AYAs with CHD to enhance their Transition Readiness. The main questions it aims to answer are:

1. Is the Get Ready with my Heart Program clinically feasible？
2. Does the Get Ready with my Heart Program improve participants' Transition Readiness?

Participants will:

1. The intervention group will receive interventions according to the Get Ready with my Heart Program, while the control group will receive standard interventions.
2. Outcome measures will be collected before the implementation of the program, and at 3 months and 6 months after the implementation.

DETAILED DESCRIPTION:
China currently has the highest number of congenital heart disease (CHD) patients in the world, placing a heavy disease burden on the country. As the number of adolescent CHD patients continues to grow, the strain on pediatric healthcare systems increases significantly, which in turn imposes a serious disease burden on families and society.

Over the past thirty years, the overall health of children and adolescents in China has greatly improved, but they are now facing new health issues and societal challenges. For example, unhealthy lifestyle behaviors are prevalent, and mental health issues are on the rise. Additionally, as treatment levels have improved, the focus of congenital heart disease care has shifted from simply improving survival rates to enhancing management throughout the entire lifecycle and overall prognosis. Effective transitional care management not only helps improve patients' self-management abilities and adherence to treatment but also reduces the socio-economic burden and enhances patients' quality of life. However, studies show that only a minority of adolescent CHD patients successfully complete this transition, highlighting the urgent need to strengthen transitional care management.

The purpose of this clinical pilot trial is to verify the feasibility and effectiveness of a management program designed to improve the transition readiness of adolescents with congenital heart disease based on the SMART model.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 12 and 21 years;
2. Diagnosed with congenital structural heart disease for at least 6 months;
3. Regularly receiving outpatient follow-up at Fudan University Children's Hospital;
4. Cognitive abilities corresponding to age, with adequate reading and comprehension skills;
5. Informed consent provided.

Exclusion Criteria:

1. Patients with physical conditions that limit participation (e.g., severe heart failure);
2. Presence of other congenital malformations (e.g., various syndromes caused by chromosomal abnormalities);
3. Patients with psychiatric disorders such as schizophrenia, intellectual disabilities, visual impairments, or other conditions that preclude participation in the study.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Self-Management and Transition to Adulthood with Rx = Treatment (STAR(x)) Questionnaire | before，3 and 6 months after intervention
  Evaluate the transition readiness levels of adolescent CHD patients using the Chinese version of Self-Management and Transition to Adulthood with Rx = Treatment (STAR(x)) . The questionnaire includes a total of 13 items across three categories: self-management (5 items), disease knowledge (3 items), and patient-doctor communication (5 items).
  It uses a 5-point Likert scale ranging from "never" to "always" or "very difficult" to "very easy," with scores assigned from 1 to 5 respectively.
  The maximum score and minimal score for the questionnaire is 65 points and 13 points, , with higher scores indicating higher levels of self-management and transition readiness.
  The questionnaire is available in both parent-reported and self-reported versions, to be filled out by the adolescent CHD patients and their primary caregivers, with consistent assessment content and scoring methods.

SECONDARY OUTCOMES:
Health-related quality of life for adolescent CHD patients | before and 6 months after intervention
  Evaluated using the Chinese version of the Pediatric Quality of Life Inventory Cardiac Module (PedsQLTM 3.0 Cardiac Module)，The PedsQL 3.0 Cardiac Module consists of 22 items across five dimensions: heart problems and symptoms (5 items), perceived physical appearance (3 items), treatment anxiety (4 items), cognitive psychological issues (5 items), and communication issues (3 items). Additionally, a medication treatment issue section (5 items) is included for children who are currently undergoing medication treatment. It uses a 5-point Likert scale ranging from 0 (Never) to 4 (Almost always). Higher scores indicate a better quality of life.
Transition skill levels for adolescent CHD patients-- General Self-Efficacy | before and 6 months after intervention
  Assessed using the General Self-Efficacy Scale (GSES) to evaluate patients' general self-efficacy and CHD disease knowledge. The Chinese version of the General Self-Efficacy Scale consists of 10 items, using a 4-point Likert scale ranging from 1 to 4. The scores of the 10 items are summed and then divided by 10 to calculate the overall scale score. A higher score indicates a higher sense of general self-efficacy.
Transition skill levels for adolescent CHD patients--Knowledge | before and 6 months after intervention
  Assessed using the Chinese version of the Leuven Knowledge Questionnaire for Congenital Heart Disease (LKQCHD) to evaluate patients' general CHD disease knowledge.The Chinese version of the LKQCHD consists of 27 items that assess the knowledge of children with congenital heart disease and their caregivers across four dimensions: (1) disease and treatment; (2) complications and prevention; (3) physical activity; (4) sexuality and genetics.
  The accuracy rate is calculated as the number of items correctly identified as "correct" divided by the total number of items, multiplied by 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No